CLINICAL TRIAL: NCT05311254
Title: A Multicenter Randomized Trial of Fosfomycin vs Ciprofloxacin for Febrile Neutropenia in Hematological Patients: Efficacy and Microbiological Safety
Brief Title: A Trial of Fosfomycin vs Ciprofloxacin for Febrile Neutropenia
Acronym: FOVOCIP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Collaborators: Instituto de Investigación Marqués de Valdecilla (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Teresa Bernal del Castillo, Principal investigator, Fundación para la Investigación Biosanitaria del Principado de Asturias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOVOCIP; 2021-000354-25 (EudraCT Number)
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, prospective, open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fosfomycin (Experimental): Drug: Fosfomycin: oral capsules containing 700 mg of calcium fosfomycin, equivalent to 500 mg of active drug.
  Interventions: Drug: Fosfomycin Calcium
- Ciprofloxacin (Active Comparator): Oral ciprofloxacin, tablets containing 500 mg of active drug.
  Interventions: Drug: Fosfomycin Calcium

INTERVENTIONS:
Drug: Fosfomycin Calcium — Oral fosfomycin, three times daily, starting from the first day of induction chemotherapy or conditioning until absolute neutrophil count >0,5x109/L.

SUMMARY:
Randomized phase 3 trial to compare efficacy and safety of oral fosfomycin versus ciprofloxacin to prevent febrile neutropenia in patients with acute leukemia or recipients of hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Multicenter, prospective, randomized, open label phase III trial to assess the efficacy and safety of oral fosfomycin vs. oral ciprofloxacin in the prevention of febrile neutropenia in patients with acute leukemia who are treated with intensive chemotherapy and/or are recipients of a hematopoietic stem cell transplant.

Non-inferiority design.

156 patients will be recruited: 78 in each arm

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand study procedures, comply with them, and provide written informed consent before any study-specific procedure.
2. Adult subjects ≥ 18 years of age with acute leukemia diagnosis who are going to receive their first intensive chemotherapy cycle or adult subjects ≥ 18 years of age who are candidates to receive a first stem cell transplant.
3. Expected neutropenia 100x109/L lasting at least seven days. In case of expected neutropenia range 100-500x109/L lasting seven days or more, at least one of the following risk factors for infection must be present:

   1. Performance status (Eastern Cooperative Oncology Group, ECOG) ≥2.
   2. Expected mucositis grade 3-4.
   3. Age ≥65 years.
   4. Comorbidity Index (HCTI) ≥3.
   5. Serum albumin< 35 g/L.
   6. Total dose of etoposide > 500 mg/m2
   7. Total dose of cytarabine > 1 g/m2
   8. Active or refractory neoplasia at the moment of stem cell transplant.
4. Performance status (Eastern Cooperative Oncology Group, ECOG) of 0 to 3.
5. Adequate organ function defined as:

   Liver: bilirubin, alkaline phosphatase, or SGOT < 3 times the upper normal limit (unless it is attributable to tumor activity).

   Renal : creatinine ≤ 250 μmol/l (2.5 mg/dL) (unless it is attributable to AML activity).
6. Life expectancy higher than 3 months.
7. Women of child-bearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of child-bearing potential and men with female partners of child-bearing potential must agree to practice 2 highly effective contraceptive measures of birth control and must agree not to become pregnant or father a child while receiving any study therapy and for at least 3 months after completing treatment.

Exclusion Criteria:

1. Hypersensitivity to fluoroquinolones or fosfomycin.
2. Treatment with broad spectrum antimicrobial therapy within 4 weeks of first study treatment.
3. Prior Intensive chemotherapy or stem cell transplant. Treatment with hydroxyurea or corticosteroids used to control white blood cell counts are permitted.
4. Fever of infectious origin or documented infection within 4 weeks of first study treatment.
5. Presence of any severe psychiatric disease or physical condition that, according to the physicians criteria, contraindicates the inclusion of the patient into the clinical trial.
6. Subjects that have participated previously in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-03-14 (Estimated); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
Febrile neutropenia of infectious origin | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Febrile neutropenia that requires antibacterial treatment.

SECONDARY OUTCOMES:
Documented infections | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Rate and type of documented infections
Use of broad spectrum antibiotics | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Index of days of antibiotics per hospitalization days. Antibiotics will be classified according the Watch/Reserve classification
Overall survival | Time from the day of randomization to the date of death, whatever the cause of death, up to 12 weeks.
Drug related adverse events | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Incidence of Adverse Events (AE), severity and type of AEs.
Evolution of resistome | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Rate of patients colonized by multidrug resistant bacteria as determined by metagenomic sequencing
Microbiome evolution | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Changes in the gut microbiome produced under both prophylactic strategies during the study period.
Microbiological safety | Immediately after the intervention until febrile neutropenia develops, neutrophil count >0,5x109/L up to 60 days maximum
  Rate of patients colonized by multidrug resistant bacteria as determined by surveillance cultures

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Bernal, MD PHD, Principal Investigator — Hospital Universitario Central Asturias
Locations (1):
- Instituto de Investigación Sanitaria del Principado de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno AF, Lavin-Alconero L, de Ugarriza PL, Blanco LS, Hernandez SC, Burgues JMB, de Miguel MI, Huerta AJG, Zarzuela MP, Boluda B, Humala K, Calabuig ML, Amigo ML, Casas MC, Del Mar Garcia-Saiz M, Verdugo AF, Dominguez JF, Bernal T. FOVOCIP study: a multicenter randomized trial of fosfomycin versus ciprofloxacin for febrile neutropenia in hematologic patients-efficacy and microbiologic safety. Trials. 2023 Oct 27;24(1):694. doi: 10.1186/s13063-023-07702-5. PMID 37891616